CLINICAL TRIAL: NCT02172326
Title: The Pharmacokinetics, Safety and Tolerability of Tiotropium in Elderly COPD Patients (Open Label, Monocenter Study).
Brief Title: Pharmacokinetic Study in Elderly Patients With Chronic Obstructive Bronchitis (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205.133
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (1):
- Tiotropium inhalation capsules (Experimental)
  Interventions: Drug: Tiotropium inhalation capsules for oral inhalation

INTERVENTIONS:
Drug: Tiotropium inhalation capsules for oral inhalation — Powder inhalation via HandiHaler®

SUMMARY:
Study to evaluate the pharmacokinetics of tiotropium following 14 days of administration (18µg once per day) in elderly COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients were required to have a diagnosis of COPD and to meet the following spirometric criteria:

  * Relatively stable, moderate to severe airway obstruction with an FEV1 ≤ 65% of predicted normal and FEV1/FVC ≤ 70%
* Patients were required to have normal renal clearance. Renal clearance will be evaluated by the determination of creatinine clearance. To qualify for this trial, the patient's measured creatinine clearance was required to be within 20% of the calculated creatinine clearance, as given by the following equations:

  * Males: Calculated Creatinine Clearance (ml/min) = [140 - Age (yrs)] x weight(kg) / 72 x serum creatinine (mg/dL)
  * Females: Calculated Creatinine Clearance (ml/min) = [140 - Age (yrs)] x weight (kg) / 85 x serum creatinine (mg/dL)
* Both male or female patients were eligible. Twelve patients ≥ 70 years old and twelve patients ≤ 50 years
* Patients were required to have a smoking history of more than ten pack-years, where a pack-year was defined as the equivalent of smoking one pack of cigarettes per day for a year
* Patients must be able to perform all specified procedures and maintain records during the study period as required in the protocol
* Patients were required to be able to inhale medication from the HandiHaler®
* Patients were required to sign an Informed Consent Form prior to participation in the trial, including any necessary prior to pre-study washout of their usual pulmonary medications

Exclusion Criteria:

* Patients with significant diseases other than COPD were excluded from participation in the trial. A significant disease was defined as a disease which in the opinion of the investigator may either have put the patient at risk because of participation in the trial or a disease which may have influenced the results of the trial or the patient's ability to participate in the trial;
* Patients with clinically significant abnormal baseline haematology, blood chemistry or urinalysis, if the abnormality defined a disease listed as an exclusion criterion;
* Patients with alanine transaminase (ALT/SGOT) > 80 IU/L or aspartate transaminase (AST/SGPT) > 80 IU/L, or bilirubin > 2.0 mg/dL or creatinine > 2.0 mg/dL were excluded from participation in the trial, regardless of the patient's clinical condition. Repeat laboratory evaluations were not conducted in these patients;
* Patients with a recent history (i.e., one year or less) of myocardial infarction (MI);
* Patients with a recent history (i.e., three years or less) of heart failure or patients with any cardiac arrhythmia requiring drug therapy;
* Patients with regular use of daytime oxygen therapy;
* Patients with known active tuberculosis;
* Patients with a history of cancer within the last five years. However, patients with treated basal cell carcinoma are allowed to participate;
* Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis;
* Patients who had undergone thoracotomy with pulmonary resection. Patients with a history of a thoracotomy for other reasons were evaluated as per exclusion criterion # 1;
* Patients who had developed an upper respiratory tract infection in six weeks prior to the Screening Visit (Visit 1) or during the baseline period;
* Patients with known hypersensitivity to anticholinergic drugs, lactose or any other components of the inhalation capsule delivery system;
* Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction;
* Patients with known narrow-angle glaucoma;
* Patients treated with cromolyn sodium or nedocromil sodium;
* Patients treated with antihistamines (H1 receptor antagonists);
* Patients using oral corticosteroid medication at unstable doses (i.e. less than six weeks on a stable dose) or at a dose in excess of the equivalent of 10 mg of prednisone per day (or 20 mg every other day);
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e. oral contraceptives, intrauterine devices, diaphragm or Norplant®);
* Patients with a history of asthma, allergic rhinitis or atopy or patients with a total blood eosinophil count ≥ 600/mm3. A repeat eosinophil count was not conducted in these patients;
* Patients with history and/or active alcohol or drug abuse.
* Patients who had taken an investigational drug within one month or six half lives (whichever was greater) prior to Screening Visit (Visit 1).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29
Dates: Start 1998-02; Primary Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
Total area under the plasma drug concentration-time curve (AUC 0-4 h) | pre-dose and 5, 20 min., 1, 2,and 4 hours after dosing on days 1, 7 and 14
Urinary excretion of tiotropium (Ae(0-4 hours)) | screening and on days 1, 7, 14, 15, 16, 20, 24, 28, 31, 35, 38
Renal clearance of tiotropium (CLren) | screening and on days 1, 7, 14, 15, 16, 20, 24, 28, 31, 35, 38
Terminal elimination half-life after the last dose | pre dose and 5, 20 min., 1, 2,and 4 hours after dosing on days 1, 7 and 14

SECONDARY OUTCOMES:
Plasma concentration of drug 5 min after inhalation (C5min) | pre dose and 5, 20 min., 1, 2,and 4 hours after dosing on days 1, 7 and 14
tmax (time of occurrence for maximum drug concentration) | pre dose and 5, 20 min., 1, 2,and 4 hours after dosing on days 1, 7 and 14
Change from baseline in FEV1 (Forced expiratory volume in one second) | Baseline, Days 1, 7 and 14
Change from baseline in FVC (Forced vital capacity) | Baseline, Days 1, 7 and 14
FEV1/FVC | Baseline, Days 1, 7 and 14
Symptom evaluation | 2 weeks
Use of salbutamol | 2 weeks
Occurrence of Adverse Events | up to day 39
Occurrence of Adverse Events | up to day 38
Changes form baseline in vital signs (pulse rate and blood pressure) | up to day 38
Changes from baseline in laboratory tests (haematology, clinical chemistry and urinalysis) | baseline, day 38
Changes from baseline in physical examination | baseline, day 38
Changes from baseline in ECG (Electrocardiogram) | baseline, day 1, 7, 14 and 38